CLINICAL TRIAL: NCT03552120
Title: The Impact of a Mindfulness-based Intervention on Opioid Use During Pregnancy: A Mixed Methods Pilot RCT
Brief Title: Serving Women Using Opioids During Pregnancy
Acronym: SWOOP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was temporarily paused due to study resources in 2019. The study was then administratively closed by the IRB due to no Continuing Review application submission prior to expiration date.
Sponsor: University of Utah (Other)
Collaborators: Mind and Life Institute, Hadley, Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_00099361
Record Dates: First submitted 2018-04-30; First posted 2018-06-11 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2020-10

CONDITIONS: Opioid Use; Pregnancy Related

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): MORE is a manualized integrative treatment strategy that targets transdiagnostic mechanisms in stress-related conditions. MORE is made up of three primary components: mindfulness training, cognitive restructuring, and savoring. Mindfulness training aims to increase attentional control to reduce cognitive bias toward negative information. Cognitive reappraisal promotes restructuring of maladaptive cognitions, which would otherwise intensify negative emotion and addictive behavior. Finally, MORE promotes savoring - mindful attention to and appreciation of pleasant events in life as a means of increasing positive emotion regulation.
  Interventions: Behavioral: MORE
- Supportive Psychotherapy (Active Comparator): Supportive psychotherapy is a form of non-directive talk therapy, which follows a Rogerian person-centered approach. The therapist's primary objectives during a session will be (1) to communicate unconditional positive regard for the participant, (2) to communicate engagement and empathic understanding, and (3) to mirror a participant's affect.
  Interventions: Behavioral: Supportive Psychotherapy

INTERVENTIONS:
Behavioral: MORE — MORE is a manualized integrative treatment strategy that targets transdiagnostic mechanisms in stress-related conditions. MORE is made up of three primary components: mindfulness training, cognitive restructuring, and savoring. Mindfulness training aims to increase attentional control to reduce cognitive bias toward negative information. Cognitive reappraisal promotes restructuring of maladaptive cognitions, which would otherwise intensify negative emotion and addictive behavior. Finally, MORE promotes savoring - mindful attention to and appreciation of pleasant events in life as a means of increasing positive emotion regulation.
  Arms: Mindfulness
Behavioral: Supportive Psychotherapy — Supportive psychotherapy is a form of non-directive talk therapy, which follows a Rogerian person-centered approach. The therapist's primary objectives during a session will be (1) to communicate unconditional positive regard for the participant, (2) to communicate engagement and empathic understanding, and (3) to mirror a participant's affect.
  Arms: Supportive Psychotherapy

SUMMARY:
The purpose of this study is to evaluate the effects of Mindfulness-Oriented Recovery Enhancement (MORE) on opioid misuse and parenting behavior among pregnant women using opioids.

Specific aims are:

AIM 1: To evaluate the preliminary efficacy of MORE, relative to a supportive counseling control condition, on primary outcomes (opioid misuse) and secondary outcomes (opioid craving, psychological distress) among pregnant women using opioids. Hypothesis: Participants who participate in MORE will demonstrate significantly greater improvements than the supportive visit control group on: opioid misuse behaviors, opioid craving, and psychological distress.

AIM 2: To test and quantify the degree to which the impact of MORE on opioid misuse is mediated by changes in cognitive, affective, and autonomic mechanisms relevant to this clinical population - including opioid attentional bias, negative emotion regulation, reward responsiveness, and physiological reactivity to infant cues. Hypothesis: The impact of MORE on craving and opioid misuse behaviors will be mediated by improvements in attentional bias toward opioid cues, negative emotion regulation and natural reward responsiveness on the emotion regulation task, and autonomic reactivity to infant cues.

AIM 3: To evaluate the impact of MORE on mothers' perceptions of their ability to parent effectively and the quality of the mother-baby relationship. Hypothesis: Participants participating in MORE will report more positive beliefs about their ability to effectively parent. Participants who participated in MORE will interact more sensitively with their newborn.

Exploratory AIM 1: To evaluate the efficacy of MORE, relative to a support group control condition, on co-regulation, as measured by an index of sympathetic nervous system functioning, among pregnant women using opioids. Hypothesis 1: Dyads in which the mother participated in MORE will demonstrate significantly greater dyadic synching of sympathetic activity as measured by respiratory sinus arrhythmia (RSA).

Exploratory AIM 2: To test and quantify the degree to which the impact of MORE on dyadic synchrony (during the Still Face Paradigm) is mediated by changes in negative emotion regulation and reward responsiveness. Hypothesis 2: The impact of MORE on dyadic synchrony will be mediated by improvements in negative emotion regulation and natural reward responsiveness as measured by an emotion regulation task.

DETAILED DESCRIPTION:
Investigators will use an embedded mixed methods design including semi-structured qualitative interviews before the intervention, after the intervention, and five months following the post-intervention assessment. For the quantitative component, investigators will use a single-blind randomized controlled design to compare within participant and between group (i.e., mindfulness vs. supportive counseling control) changes in opioid misuse and craving as well as the quality of the mother-baby relationship. Psychophysiology will be used to assess the neurocognitive and autonomic mediators of treatment effects.

After determining eligibility, participants will be consented by the Principal Investigator or a research assistant. During the consent visit, individuals will also participate in a structured psychiatric interview, an opioid misuse assessment, and self-report measures. During a second visit, individuals will complete a psychophysiological protocol. All assessments will be conducted in the participant's home, at the University of Utah College of Social Work in Dr. Eric Garland's lab and the Bridge Training Clinic, or at the participant's physician's office or substance use treatment facility.

Psychiatric interview and opioid misuse assessment: Mini-International Neuropsychiatric Interview 6.0 and Addiction Behaviors Checklist.

Self report measures: The following validated questionnaires will be administered: Brief Pain Inventory; Current Opioid Misuse Measure; Opioid Craving Visual Analogue Scale; Depression Anxiety Stress Scale; Five Facet Mindfulness Questionnaire; Cognitive Emotion Regulation Questionnaire; Brief Savoring Beliefs Inventory; Attention to Positive and Negative Information Scale; Multidimensional Assessment of Interoceptive Ability; Coping Strategies Questionnaire; Ways of Savoring Checklist; Maternal Antenatal Attachment Scale; the Parenting Stress Index; the Edinburgh Postnatal Depression Scale; the Interpersonal Mindfulness in Parenting Scale - Infant Version; the Parental Evaluation Scale; the Self-Compassion Scale; Brief Child Abuse Potential Inventory.

Psychophysiological protocol:

To assess for attentional bias to opioid-related and natural reward cues, investigators will employ a dot probe task to measure reaction times (RTs) to target probes replacing neutral photos compared with RTs to probes replacing opioid-related photos (e.g., pills, pill bottles) and natural reward photos (e.g., smiling babies, food). Reward and neutral photos will be selected from the International Affective Picture System and opioid-related photos will be taken from media libraries on the internet. Equal proportions neutral/reward, and neutral/opioid stimuli will be presented. Each pair of stimuli will be presented for 50 ms, 200 ms, or 2000 ms on either side of a fixation cross. A target probe will replace one of the photos after a 50 ms interstimulus interval (ISI). Cue/target probe position and presentation duration will be pseudo-randomized and counterbalanced. RTs and accuracy will be analyzed.

To measure emotion regulation and natural reward responsiveness, investigators will use a well-validated emotion regulation task in which a trial will be composed of six parts. First, a fixation cross will appear for 3-7 seconds. Then, a negative or positive emotional image will appear for 2 seconds to elicit an emotional response. Next, a semi-transparent instruction ("Reappraise," "Savor," or "Look") will appear below the image for 2 seconds. A research assistant will instruct the participant before the task begins to down-regulate emotion on negative affect trials and up-regulate emotion on positive affect trials. Next, the image will appear alone on the screen for 6 seconds during which time participants will implement the instructed strategy. Negative (e.g., angry faces, violent scenes) and positive images (e.g., smiling persons, nature scenes) will be selected from the IAPS (M valence: neg=2.7; pos=7.0) and equated on mean arousal (neg=5.3; pos=5.3). At the end of the trial, participants will rate their affective response. Twelve trials of each event type will be randomly presented over four 6-minute runs.

Psychophysiological responses (HR, HRV, SCR, RSA) during the dot probe and emotion regulation tasks will be collected via ECG monitor, respiration belt, and Electrodermal Activity Amplifier, and assessed with a BIOPAC psychophysiological data acquisition unit during the dot probe and emotion regulation tasks. R-waves and SCRs will be inspected for artifacts and corrected according to established guidelines. HR, and SCR cue-responses will be calculated by subtracting mean values prior to cue onset from maxima during cue exposure as well as from each 25ms epoch during photo presentation. Time domain and spectral HRV analyses will be computed with FFT and autoregressive algorithms. HRV during task blocks will be compared to 5-min baseline and recovery periods.

Infant Cry Stimulus: Participants will be asked to watch a video during which an infant is playing and smiling and then begins to cry. investigators will measure participants' physiological reactions to watching the video. In the first three minutes of the video, participants will watch a tranquil seascape scene during which baseline physiology will be measured. Then, they will watch 35-seconds or the infant playing with her mother. Following this interaction on the video, the mother stops playing with the infant who immediately begins crying. She cries for 2.5 minutes. investigators refer to this segment as the infant cry segment. This exact stimulus has been used in previous research and moderate increases in heart rate and decreases in respiratory sinus arrhythmia (RSA) were observed, indicative of a moderate response to stress.

After completing the pre-assessments, individuals will be randomly assigned to participate in 8 weeks of MORE or 8 weeks of supportive counseling visits using a validated control condition protocol. MORE consists of three components: mindfulness, reappraisal, and savoring. This intervention was developed specifically for individuals using opioids. The supportive counseling control will be matched for time and attention from a professional. In this condition, the therapist will actively listen and validate the participant's experiences, but will not provide any coping skills training. The interventions will be delivered in individual sessions either in the participant's home, at the College of Social Work Bridge Training Clinic, or at the participant's medical clinic or substance use facility. During the last session, the therapist will conduct a semi-structured interview focused on the participant's experience of the intervention. During the last session, the therapist will conduct a semi-structured interview focused on the participant's experience of the intervention. Importantly, these sessions will be audio recorded and a random selection will be assessed for treatment fidelity. The recordings will also be transcribed and analyzed for themes.

After eight weeks of participating in MORE or supportive counseling, participants will complete two post-treatment assessments mirroring the initial assessments. Part one will consist of the opioid misuse assessment and self-report measures. Part two will consist of the psychophysiological protocol.

The research assistants and Dr. Conradt will be notified via theradoc (email) when patient is admitted to the hospital and is in labor. Investigators will collect the placenta within 4 hours of delivery using our established methods of placenta collection from IRB 81198 (BABY study). Twenty-four hours after delivery we will conduct the standardized newborn neurobehavioral assessment (NNNS) which is currently being used in our NIH-funded research and in IRB 81198 (BABY study).

When the child is five months old, the participant will return for a follow-up visit. This assessment will include the opioid misuse assessment, a mother-baby interaction assessment, and the Still Face Paradigm. Importantly, the mother-baby interaction and Still Face Paradigm will be filmed to be assessed by a second research assistant. During the mother-baby interaction assessment, a research assistant (blind to treatment condition) will behaviorally code the mother-baby interaction while viewing this interaction from behind a one-way mirror. During the interaction, research assistants will code discrete infant behaviors (e.g. the amount of time the infant is crying during the interaction) and discrete mother behaviors (e.g., the amount of time mother spends interacting insensitively with the infant).

During the Still Face Paradigm, the participant is instructed to interact normally with her baby for two minutes, to then stop interacting with her baby for two minutes, and to then resume interacting with her baby for two minutes. During this assessment, mother and baby will be both be fit with ECG electrodes to measure heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant
* Taking opioids (prescription opioids, methadone, suboxone, heroin, kratom, etc.)
* Fluent in English

Exclusion Criteria:

* Past experiences with mindfulness-based stress reduction, mindfulness-based relapse prevention, mindfulness-based cognitive therapy
* Active suicidality
* Active psychosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Current Opioid Misuse Measure | 10 weeks
  The Current Opioid Misuse Measure misuse (COMM; α = .83) is a 17-item scale developed to help physicians identify patients misusing their prescribed opioids. Examples of items include: "In the past 30 days, how often have you needed to take pain medications belonging to someone else?" and, "In the past 30 days, how often have you used your pain medicine for symptoms other than for pain (e.g., to help your sleep, improve your mood, or relieve stress)?"
Brief Child Abuse Potential Inventory | 10 weeks
  The Brief Child Abuse Potential Inventory (B-CAP; α = .89) was developed from the Child Abuse Potential Inventory to identify in a briefer time period individuals at risk for committing child abuse. The B-CAP is a 24-item self-report scale with disagree and agree responses. Items include "Children should never disobey", "Children should be quiet and listen", and "A child needs very strict rules."

SECONDARY OUTCOMES:
Opioid Craving Visual Analog Scale | 10 weeks
  Opioid craving will be measured using seven questions with a visual analog scale from 0 to 100 (opioid visual analog scale). Questions include "In the past 24 hours, how strong of an urge did you have to take more opioid medication than prescribed?" and "In the past 24 hours, how often have you found yourself thinking about the next opioid dose?"
Depression, Anxiety and Stress Scale | 10 weeks
  Psychological distress will be measured using the composite score of a 21-item Depression, Anxiety, and Stress Scale (DASS-12; α = .93). Some items include "I found myself getting upset by quite trivial things," "I felt I had nothing to look forward to," and "I felt scared without any good reason." Responses range from 0, Did not apply to me at all, to 3, Applied to me very much, or most of the time.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Priddy, MSW, Principal Investigator — University of Utah
Locations (1):
- The University of Utah, Salt Lake City, Utah, United States